CLINICAL TRIAL: NCT00444535
Title: A Phase II, Open-Label Study of the Clinical Activity, Safety, and Tolerability of Lapatinib in Combination With Bevacizumab in Subjects With Advanced or Metastatic ErbB2-Overexpressing Breast Cancer
Brief Title: Lapatinib and Bevacizumab for Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Masking: None | Purpose: Treatment
Other Study IDs: EGF103890; CLAP016A2201 (Other: Novartis)
Record Dates: First submitted 2007-03-06; First posted 2007-03-08 (Estimated); Results first posted 2009-08-20 (Estimated); Last update posted 2021-10-25 (Actual); Status verified 2021-09

CONDITIONS: Neoplasms, Breast
Keywords: VEGF; Tyrosine kinase; ErbB2; Her2-neu; metastatic breast cancer; EGFR; ErbB1; bevacizumab; lapatinib; breast carcinoma; breast cancer; breast lump; breast cancer positive for human epidermal growth factor receptor 2 (HER2); HER2 positive metastatic breast cancer; breast cancer progression; estrogen-receptor (ER) positive(+) breast cancer; Paget's disease
MeSH Terms: conditions — Breast Neoplasms; Osteitis Deformans | interventions — Lapatinib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oral lapatinib tablets in combination with IV bevacizumab (Experimental): 1500 mg oral lapatinib (once daily) plus 10 mg/kg intravenous bevacizumab (every two weeks)
  Interventions: Drug: lapatinib; Drug: bevacizumab

INTERVENTIONS:
Drug: lapatinib — 1500 mg oral lapatinib (once daily)
  Other Names: Tykerb/Tyverb
Drug: bevacizumab — 10 mg/kg intravenous bevacizumab (every two weeks)

SUMMARY:
This study will examine the efficacy and safety of lapatinib and bevacizumab in patients with ErbB2-overexpressing breast cancer.

ELIGIBILITY:
Inclusion criteria:

* Females that are at least 18 years of age.
* Women of childbearing potential must have a negative serum pregnancy test at screening.
* Documented evidence of HER2-overexpressing unresectable or metastatic breast cancer. Disease may/may not have been treated in metastatic setting.
* Subjects are permitted (but not required) to have previously-treated brain metastases that are stable and asymptomatic.
* Adequate hepatic, renal and cardiac function
* ECOG score 0-1 and a life expectancy of at least 12 weeks.
* Able to swallow oral medication
* Signed informed consent

Exclusion criteria:

* Pregnancy
* Unstable or symptomatic CNS metastases
* Major surgery within 28 days of enrollment (minor surgery within 7 days).
* Prior anti-cancer treatment within 14 days of enrollment, or unresolved treatment-related toxicities.
* A serious non-healing wound, ulcer, or bone fracture at baseline.
* Class II, III or IV heart failure as defined by the NYHA functional classification system
* History of significant vascular disease, arterial thrombosis, unstable INR, hypertensive crisis, or uncontrolled hypertension.
* History of myocardial infarction, stenting procedure, or angioplasty within 6 months of enrollment.
* History of abdominal fistulae, gastrointestinal perforation, or intra-abdominal abscess within 6 months of enrollment.
* History of malabsorption syndrome, ulcerative colitis, or bowel obstruction.
* Proteinuria
* Requires concurrent anti-cancer treatment or investigational treatment.
* Known hypersensitivity to either study medication
* Received investigational treatment within 28 days or 5 half-lives, whichever is longer
* Concurrent disease or circumstances that would lead the investigator would consider the subject an inappropriate candidate for the study
* Requires medication that has been excluded during study participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-02-27 (Actual); Primary Completion 2008-07-22 (Actual); Study Completion 2020-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- United States (9):
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Hollywood, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Basking Ridge, New York
  - Novartis Investigative Site, Commack, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Rockville Centre, New York
  - Novartis Investigative Site, Sleepy Hollow, New York

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- [Background] Rugo HS, Chien AJ, Franco SX, Stopeck AT, Glencer A, Lahiri S, Arbushites MC, Scott J, Park JW, Hudis C, Nulsen B, Dickler MN. A phase II study of lapatinib and bevacizumab as treatment for HER2-overexpressing metastatic breast cancer. Breast Cancer Res Treat. 2012 Jul;134(1):13-20. doi: 10.1007/s10549-011-1918-z. Epub 2011 Dec 24. PMID 22198412

RESULTS

PARTICIPANT FLOW:
Groups:
- Lapatinib + Bevacizumab: Lapatinib (1500 mg once daily taken orally) and bevacizumab (10 mg/kg intravenously [IV] every two weeks)
Period: Overall Study
Arm/Group | Lapatinib + Bevacizumab
Started | 52
Completed | 39
Not Completed | 13
Not completed — Withdrawal by Subject | 5
Not completed — Physician Decision | 5
Not completed — progressive disease | 1
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Lapatinib + Bevacizumab
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White/Caucasian/European Heritage | 42
  African American/African Heritage | 7
  Asian | 2
  Asian and White | 1

OUTCOME MEASURES:

1. Primary Outcome: Investigator-evaluated Crude Progression-free Survival Rate After 12 Weeks of Study Treatment
Description: The PFS rate is defined as the percentage of subjects who have shown no evidence of disease progression or death from any cause following 12 weeks of treatment. Disease progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
  Since there is no independent reviewer, only the investigator response was reported.
Time Frame: up to week 12
Population: Intent-to-Treat (ITT) Population: all enrolled participants, regardless of whether or not they received any study medication
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib + Bevacizumab
Number analyzed (Participants) | 52
Participants
  No disease progression by Week 12 | 36
  Disease progression or death by Week 12 | 16
Statistical Analysis 1: Comparison: Lapatinib + Bevacizumab; Test type: Other — Clopper-Pearson exact test (binomial); Exact binomial procedure = 69.2, 95% CI [54.9 to 81.3]

2. Secondary Outcome: Overall Tumor Response - Best Response Per Investigator Assessment (RECIST)
Description: Overall Tumor Response - Best Response per Investigator Assessment Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by image including CT, MRI or bone scan: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
  For each subject, the best tumor response during the study was considered to be the 'Overall Tumor Response' per the Response Evaluation Criteria in Solid Tumors (RECIST).
Time Frame: This endpoint was defined in the original protocol but was cancelled per Amendment 3, which was implemented Nov 2015. The timeframe therefore is from treatment start to Nov 2015, with a maximum timeframe of approx. 8.7 years.
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib + Bevacizumab
Number analyzed (Participants) | 52
Participants
  Complete response | 0
  Partial response | 7
  Stable disease | 26
  Progressive Disease | 11
  Unknown | 8

3. Secondary Outcome: Overall Tumor Response Rate Per Investigator Assessment (RECIST)
Description: Overall Tumor Response Rate is defined as the percentage of subjects achieving either a confirmed complete (CR) or partial (PR) tumor response by investigator and per the Response Evaluation Criteria in Solid Tumors (RECIST). For each subject, the best tumor response during the study are considered the 'Overall Tumor Response.' Subjects with unknown or missing response are treated as non-responders; i.e. they are included in the denominator when calculating the percentage.
Time Frame: as for outcome 2
Population: ITT Population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lapatinib + Bevacizumab
Number analyzed (Participants) | 52
Percentage of participants | 13.5 [5.6 to 25.8]

4. Secondary Outcome: Investigator-Assessed Clinical Benefit Response Rate (%) (RECIST)
Description: Clinical Benefit Rate is defined as the percentage of subjects with evidence of confirmed complete or partial tumor responses at any time or stable disease for at least 24 weeks per the Response Evaluation Criteria in Solid Tumors (RECIST). Subjects with unknown or missing response are treated as non-responders (i.e. not Complete response (CR), Partial response (PR) or Stable Disease (SD)).
Time Frame: as for outcome 2
Population: ITT Population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lapatinib + Bevacizumab
Number analyzed (Participants) | 52
Percentage of participants | 38.5 [15.4 to 59.2]

5. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) = time from treatment start date until the first documented sign of disease progression, as defined by the investigator, or death due to any cause. For participants who did not progress or die at the time of reporting, PFS data were censored at the time of the last radiological assessment.
Time Frame: as for outcome 2
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib + Bevacizumab
Number analyzed (Participants) | 52
Participants
  Progressed or Died (event) | 39
  Censored, Follow-up ended | 13

6. Secondary Outcome: Progression-free Survival - Kaplan-Meier Estimates for Progression-free Survival (Weeks) - Median
Description: Progression-free survival (PFS) = time from treatment start date until the first documented sign of disease progression, as defined by the investigator, or death due to any cause. For participants who did not progress or die at the time of reporting, PFS data were censored at the time of the last radiological assessment. Greenwood's formula was used to calculate the standard error of the estimates from the Kaplan-Meier curve.
Time Frame: as for outcome 2
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lapatinib + Bevacizumab
Number analyzed (Participants) | 52
weeks | 24.7 [20.9 to 33.1]

7. Secondary Outcome: Progression-free Survival - Kaplan-Meier Estimates for Progression-free Survival (Weeks) - 1st and 3rd Quartile
Description: as for outcome 6
Time Frame: as for outcome 2
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | Lapatinib + Bevacizumab
Number analyzed (Participants) | 52
weeks
  Estimates for progression-free survival 1st Quartile (weeks) | 12.9 [6.1 to 21.4]
  Estimates for progression-free survival 3rd Quartile (weeks) | 35.6 [31.1 to 61.3]

ADVERSE EVENTS:
Time Frame: Adverse events are reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of 634 weeks (12.2 yrs).
Groups:
- Lapatinib + Bevacizumab: Lapatinib + Bevacizumab
Arm/Group | Lapatinib + Bevacizumab
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 13/52
Other Adverse Events (participants affected / at risk) | 52/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib + Bevacizumab (N=52)
Anaemia (Blood and lymphatic system disorders) | 1
Blood loss anaemia (Blood and lymphatic system disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Gastric haemorrhage (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Pyrexia (General disorders) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Ejection fraction decreased (Investigations) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Hydronephrosis (Renal and urinary disorders) | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib + Bevacizumab (N=52)
Vision blurred (Eye disorders) | 4
Abdominal distension (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 10
Diarrhoea (Gastrointestinal disorders) | 41
Dry mouth (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 4
Gingival bleeding (Gastrointestinal disorders) | 3
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 3
Haemorrhoids (Gastrointestinal disorders) | 4
Mouth ulceration (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 25
Vomiting (Gastrointestinal disorders) | 17
Asthenia (General disorders) | 3
Chills (General disorders) | 3
Fatigue (General disorders) | 32
Mucosal inflammation (General disorders) | 10
Pain (General disorders) | 3
Pyrexia (General disorders) | 3
Nasopharyngitis (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 4
Contusion (Injury, poisoning and procedural complications) | 3
Fall (Injury, poisoning and procedural complications) | 3
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 3
Weight decreased (Investigations) | 6
Decreased appetite (Metabolism and nutrition disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 12
Back pain (Musculoskeletal and connective tissue disorders) | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 24
Memory impairment (Nervous system disorders) | 3
Neuropathy peripheral (Nervous system disorders) | 3
Paraesthesia (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 5
Anxiety (Psychiatric disorders) | 6
Depression (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 6
Proteinuria (Renal and urinary disorders) | 6
Vulvovaginal dryness (Reproductive system and breast disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 21
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 6
Nail disorder (Skin and subcutaneous tissue disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 32
Hypertension (Vascular disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.